CLINICAL TRIAL: NCT04922632
Title: Data-driven Approaches to Healthcare Provider Resilience & Burnout During COVID-19
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding was exhausted
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00106079
Record Dates: First submitted 2021-06-08; First posted 2021-06-10 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Burnout, Professional; Exhaustion, Caregiver; Covid19
MeSH Terms: conditions — Burnout, Professional; Caregiver Burden; COVID-19 | interventions — Meditation; Therapeutics

STUDY DESIGN:
Intervention Model Description: A 4-year, multi-site, four-arm parallel-group randomized clinical trial (RCT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Transcendental Medication (TM) (Experimental): Transcendental Meditation (TM): a mind-body program that allows the participant to experience progressively quieter, less excited states of mental activity, with growing experience of restful alertness in mind and body.
  Interventions: Behavioral: Transcendental Meditation (TM)
- Experience Resolution Methodology (ERM) (Experimental): Experience Resolution Methodology (ERM): is a specific, protocolized coaching method that aims to maximize an individual's performance, professional development and well-being by recognizing and resolving subjective stress associated with specific situations, circumstances, events or experiences.
  Interventions: Behavioral: Experience Resolution Methodology (ERM)
- TM+ERM (Experimental): Transcendental Meditation (TM) and Experience Resolution Methodology (ERM): an integrative method using both TM and ERM coaching with ERM with the aim of achieving an overall restful, alertness in mind and body and maximizing performance, professional development and well-being.
  Interventions: Behavioral: Transcendental Meditation (TM) and Experience Resolution Methodology (ERM)
- Treatment As Usual (TAU) (Active Comparator): Treatment As Usual (TAU): is the existing Duke Health & Well-being services, such as the availability of acupuncture, integrative health coaching, integrative nutrition and weight management, personal exercise training, massage therapy, yoga therapy, mindfulness-based stress reduction (MBSR), experiencing mindfulness, group fitness classes, gentle yoga, or chair yoga, as well as additional resources such as Personal Assistance Services (PAS).
  Interventions: Behavioral: Treatment As Usual (TAU)

INTERVENTIONS:
Behavioral: Transcendental Meditation (TM) — TM is a mind-body program that allows the participant to experience progressively quieter, less excited states of mental activity, with growing experience of restful alertness in mind and body.
  Arms: Transcendental Medication (TM)
Behavioral: Experience Resolution Methodology (ERM) — ERM is a specific, protocolized coaching method that aims to maximize an individual's performance, professional development and well-being by recognizing and resolving subjective stress associated with specific situations, circumstances, events or experiences.
  Arms: Experience Resolution Methodology (ERM)
Behavioral: Transcendental Meditation (TM) and Experience Resolution Methodology (ERM) — TM + ERM is an integrative method using both TM and ERM coaching with ERM with the aim of achieving an overall restful, alertness in mind and body and maximizing performance, professional development and well-being.
  Arms: TM+ERM
Behavioral: Treatment As Usual (TAU) — TAU is the existing Duke Health & Well-being services, such as the availability of acupuncture, integrative health coaching, integrative nutrition and weight management, personal exercise training, massage therapy, yoga therapy, mindfulness-based stress reduction (MBSR), experiencing mindfulness, group fitness classes, gentle yoga, or chair yoga, as well as additional resources such as Personal Assistance Services (PAS).
  Arms: Treatment As Usual (TAU)

SUMMARY:
The United States is battling dual pandemics: healthcare provider (HCP) exhaustion and COVID-19. The COVID-19 pandemic death toll has surpassed 595,000 and continues to climb as the worldwide outbreak continues. Moreover, we have yet to understand the health impacts of "long-COVID". As evidenced by the national burnout epidemic in HCPs, persistent workplace stress not only impacts personal provider wellbeing, but also influences effective practice and patient outcomes.

To address this need, we propose a 4-year, multi-site, four-arm parallel-group randomized clinical trial (RCT) comparing 2 non-pharmacological interventions: Transcendental Meditation (TM) and Experience Resolution Methodology (ERM) to Treatment as Usual (TAU).

Participation in this study lasts up to 24 months for enrolled participants and is considered minimal risks.

DETAILED DESCRIPTION:
The United States is battling dual pandemics: healthcare provider (HCP) exhaustion and COVID-19. The COVID-19 pandemic death toll has surpassed 595,000 and continues to climb as the worldwide outbreak continues. Moreover, we have yet to understand the health impacts of "long-COVID". Taxed with an overloaded healthcare system, longer shifts, disrupted work-life balance, and the responsibility to uphold biosecurity with limited personal protective equipment (PPE), frontline HCPs are experiencing unprecedented levels of distress. A major and shared anxiety among HCPs is the fear of propagating the disease to their coworkers and their families. As evidenced by the national burnout epidemic in HCPs, persistent workplace stress not only impacts personal provider wellbeing, but also influences effective practice and patient outcomes.

National institutes, such as the Joint Commission, are calling for the prioritization of healthcare workforce resilience in an effort to protect against rapid turnover, medical errors and suboptimal patient care. Resilience is defined as the "ability to respond to stress in a healthy, adaptive way, such that goals are met with minimal psychologic and physical cost". However, the major obstacle to systematically addressing HCPs burnout and building a resilience-based workforce is the sparsity of data on qualitative, physiologic, and biological predictors of resilience and evidence-based preventative, diagnostic, and treatment strategies. At this point, most health care institutions, if they are addressing burnout and resilience at all, offer a form of executive coaching. However, there is limited systematic evidence to support benefit.

To address this need, we propose a 4-year, multi-site, four-arm parallel-group randomized clinical trial (RCT) that will be operationalized via three distinct aims:

* Aim 1: To assess the efficacy of 1) Transcendental Meditation® (TM®) versus Treatment as Usual (TAU), 2) a form of coaching termed Experience Resolution Methodology (ERM) versus TAU, and 3) TM plus ERM versus TAU in increasing resilience and reducing burnout syndrome in HCPs.
* Aim 2: To characterize the biometric, immunologic, and neuro-functional characteristics of HCPs' resilience and burnout.
* Aim 3: To develop a medical predictive model and a composite resilience and burnout index.

For this study, the term "health care provider" (HCP) will be all inclusive of any individual working in a health care setting with patient-facing responsibilities in addition to physician and physician trainees.

ELIGIBILITY:
Inclusion Criteria:

1. Full-time HCPs
2. A score of >= 5 on the Subjective Units of Distress Scale (SUDS) at baseline visit.
3. Willingness to address burnout symptoms by non-pharmacological means.
4. Willingness to wear the provided wearable device (e.g., Apple, Empatica, and/or eSense) at the designated study visits and/or determined coaching sessions, as well as wear an Apple device, if eligible to receive an Apple watch, from baseline for the duration of the study (up to 24 months).
5. Willingness to download the PatternHealth app on personal device.

Exclusion Criteria:

1. Addition or change in dosage of psychotropic medications, beta-blockers, or anti-epileptic medications within the last 2 months
2. HCPs may re-present for screening again after 2 months has passed since their last change in the medication categories listed that previously excluded them for re-evaluation for study eligibility.
3. Current suicidal or homicidal ideation at the time of screening, as defined by the C-SSRS.
4. Prior instruction in the Transcendental Meditation (TM) technique by a certified instructor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2023-03-12 (Actual); Study Completion 2023-03-12 (Actual)

PRIMARY OUTCOMES:
Change in resilience as measured by the Connor-Davidson Resilience Scale-25 | Baseline to 3 months
  The Connor-Davidson Resilience scale (CD-RISC) comprises of 25 items, each rated on a 5-point scale (0-4), with higher scores reflecting greater resilience

SECONDARY OUTCOMES:
Change in burnout as measured by the Maslach Burnout Inventory (MBI). | Baseline to 3 months
  The MBI consists of 3 scales to assess emotional exhaustion, depersonalization, and personal accomplishment with higher scores reflecting greater burnout. The MBI is composed of 22 items, each rated on a scale of 0 to 6, 0 being equivalent to "never" and 6 being equivalent to "every day." The lower scores reflect greater burnout.
Change in depression as measured by the Patient Health Questionnaire-9 (PHQ-9). | Baseline to 3 months
  The PHQ-9 is a 9 question survey that rates responses on a scale of 0 to 3, 0 being equivalent to "not at all" and 3 equivalent to "nearly every day". The higher scores reflect greater depression in an individual.
Change in psychological distress as measured by the Subject Units of Distress Scales (SUDS). | Baseline to 3 months
  The Subjective Units of Distress Scale (SUDS) is a 0 to 10 scale, 0 being "totally relaxed" and 10 being "highest/distress/fear/anxiety/discomfort that you have ever felt". The SUDS measures subjective intensity of disturbance or distress. The higher the score the great the individual's psychological distress.
Change in quality of life as measured by the Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF). | Baseline to 3 months
  The Q-LES-Q-SF is an assessment that measures the degree of enjoyment and satisfaction experienced by individuals in various areas of daily functioning. It is a 16 item assessment on a scale of 1 to 5, 1 being equivalent to "very poor" and 5 being equivalent to "very good." The higher scores reflect increased perceived quality of life.
Change in PTSD symptom severity as measured by the Post-Traumatic Stress Disorder (PTSD) checklist-5 (PCL-5). | Baseline to 3 months
  The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD rated on a scale of 0 to 4, 0 being "not at all" and 4 "extremely." The higher scores reflect greater PTSD.
Change in sleep as measured by the Insomnia Severity Index (ISI). | Baseline to 3 months
  The ISI is a patient-reported outcome that assesses the individual's sleep patterns over the past 2 weeks. The ISI is a 7 item questionnaire on a scale of 0 to 4, 0 being "none" and 4 being "very severe". The higher score indicates worse sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Sangeeta Joshi, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data, post analysis may be shared with other researchers at scientific meetings and published within scientific journals.

DOCUMENTS (1):
  • Informed Consent Form (2023-03-08): https://cdn.clinicaltrials.gov/large-docs/32/NCT04922632/ICF_000.pdf